CLINICAL TRIAL: NCT01757964
Title: Bacteriotherapy in Pediatric Inflammatory Bowel Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: David Suskind (Other)
Collaborators: Seattle Children's Hospital (Other)
Responsible Party: Sponsor-Investigator, David Suskind, Associate Professor of Pediatrics, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14267
Record Dates: First submitted 2012-12-22; First posted 2012-12-31 (Estimated); Results first posted 2016-05-25 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis; CD
Keywords: Crohns Disease; Ulcerative Colitis; Inflammatory Bowel Disease; IBD
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bacteriotherapy (Experimental): Study stool recipient's will receive approximately 30 grams of processed donor stool through a tube into their stomach for the transplant.
  Interventions: Biological: Bacteriotherapy

INTERVENTIONS:
Biological: Bacteriotherapy

SUMMARY:
In this study, the investigators want to see if Bacteriotherapy (also referred to as stool transplantation) improves the symptoms and decreases inflammation in children with Inflammatory Bowel Disease (IBD). Examples of IBD are Crohn's Disease and Ulcerative Colitis. Additionally, researchers want to learn whether this experimental therapy delays the need for starting additional medications to treat pediatric IBD.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 12-21 years old with a diagnosis of mild to moderate Ulcerative Colitis or Crohn's Disease
* Willing parent to donate stool for the transplant

Exclusion Criteria:

* Severe Disease
* History of intra-abdominal abscess, intra-abdominal fistula or stricturing
* History of other systemic diseases
* The patient has received TNF inhibitors to treat their IBD within two months of transplant

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2012-12; Primary Completion 2013-10 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

REFERENCES:
- [Result] Suskind DL, Brittnacher MJ, Wahbeh G, Shaffer ML, Hayden HS, Qin X, Singh N, Damman CJ, Hager KR, Nielson H, Miller SI. Fecal microbial transplant effect on clinical outcomes and fecal microbiome in active Crohn's disease. Inflamm Bowel Dis. 2015 Mar;21(3):556-63. doi: 10.1097/MIB.0000000000000307. PMID 25647155
- [Result] Suskind DL, Singh N, Nielson H, Wahbeh G. Fecal microbial transplant via nasogastric tube for active pediatric ulcerative colitis. J Pediatr Gastroenterol Nutr. 2015 Jan;60(1):27-9. doi: 10.1097/MPG.0000000000000544. PMID 25162366

RESULTS

PARTICIPANT FLOW:
Groups:
- Bacteriotherapy: Crohn's Disease; Bacteriotherapy: Ulcerative Colitis: Initial evaluation: Study subject recipient had laboratory tests Stool Transplantation: Study subject recipients received premedication prior to fecal transplant, which included rifaximin. Study subject recipients also receive Omeprazole (1mg/kg orally) on the day before and morning of procedure. Transplant recipient also MiraLAX for 2 days prior to FMT. For the FMT, a nasogastric (NG) tube was placed. Approximately 30g of donor stool was mixed with 100ml of normal saline and blenderized until a homogenous texture was achieved Post Transplantation follow-up: Study subject recipients were called 2 days after transplantation. Study subject recipients had clinical follow-up at 2 weeks, 6 weeks and 12 weeks. Standardized questionnaires, PUCAI, were completed during each study visit.
Period: Overall Study
Arm/Group | Bacteriotherapy: Crohn's Disease | Bacteriotherapy: Ulcerative Colitis
Started | 9 | 4
Completed | 9 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bacteriotherapy: Crohn's Disease | Bacteriotherapy: Ulcerative Colitis | Total
Number analyzed (Participants) | 9 | 4 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 4 | 9
  Between 18 and 65 years | 4 | 0 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Responded to Stool Translplantation By 2 Weeks as Determined by Pediatric Ulcerative Colitis Activity Index (PUCAI)/Pediatric Crohn's Disease Activity Index (PCDAI) Scoring
Description: The primary outcome measure is based on estimating the responder rate. This is defined as the proportion of patients with response to therapy by a drop of 10 or more points in PUCAI/PCDAI scoring. PUCAI/PCDAI are validated activity indexes for pediatric Ulcerative colitis and Crohn's disease, respectively. PUCAI scoring ranges from 0 to 85, with disease remission less than 10, mild disease activity between 10 - 35, moderate disease activity from 35 - 65, and severe disease activity above 65. PCDAI scoring ranges from 0 to 100; with remission being less than 10, mild disease from 10 to 30, and moderate to severe disease greater than 30.
Time Frame: 2 weeks
Measure: Number; unit: participants
Groups:
- Bacteriotherapy: Study stool recipient's will receive approximately 30 grams of processed donor stool through a tube into their stomach for the transplant.
  Bacteriotherapy
Arm/Group | Bacteriotherapy
Number analyzed (Participants) | 13
participants | 13

ADVERSE EVENTS:
Groups:
- Bacteriotherapy: Initial evaluation: Study subject recipient had laboratory tests Stool Transplantation: Study subject recipients received premedication prior to fecal transplant, which included rifaximin. Study subject recipients also receive Omeprazole (1mg/kg orally) on the day before and morning of procedure. Transplant recipient also MiraLAX for 2 days prior to FMT. For the FMT, a nasogastric (NG) tube was placed. Approximately 30g of donor stool was mixed with 100ml of normal saline and blenderized until a homogenous texture was achieved Post Transplantation follow-up: Study subject recipients were called 2 days after transplantation. Study subject recipients had clinical follow-up at 2 weeks, 6 weeks and 12 weeks. Standardized questionnaires, PUCAI, were completed during each study visit.
Arm/Group | Bacteriotherapy
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 6/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bacteriotherapy (N=13)
Abdominal pain (Gastrointestinal disorders) | 5 (5) — Mild(4/5);moderate(1/5); all self resolving.
Mild bloating (Gastrointestinal disorders) | 6 (6) — Mild self resolving.
Diarrhea (Gastrointestinal disorders) | 4 (4) — Mild self resolving.
Flatulence (Gastrointestinal disorders) | 2 (2)
Rhinorrhea (Ear and labyrinth disorders) | 1 (1) — Related to nasogastric tube placement. Self resolved.
Sore throat (Gastrointestinal disorders) | 2 (2) — Self resolving. Related to Nasogastric tube placement.
Nasal congestion (General disorders) | 1 (1) — mild self resolving related to the nasogastric tube placement
Vomiting (Gastrointestinal disorders) | 2 (2) — Episodes occurred greater than 4 hours after FMT. One related to 3 hour car ride after FMT the other associated with eating a large greasy meal after FMT.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No